CLINICAL TRIAL: NCT02001753
Title: Impact of Cardiac Magnetic Resonance Imaging on Endothelial Function in Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xiang Guang-da (Other)
Responsible Party: Sponsor-Investigator, Xiang Guang-da, Director of Endocrinology, Wuhan General Hospital, Wuhan General Hospital of Guangzhou Military Command
Organization: Wuhan General Hospital of Guangzhou Military Command (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Wze20130100
Record Dates: First submitted 2013-11-23; First posted 2013-12-05 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-04

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CMR group (Experimental): Endothelial function, oxidative stress and inflammation were measured before and after CMR.
  Interventions: Device: CMR
- Placebo group (Placebo Comparator): The subjects keep supine position the MR machine as same time as experimental group when the MR machine is power off. The endothelial function, oxidative stress and inflammation were measured before and after this procedure". This group is called the non-CMR group or sham CMR group.
  Interventions: Device: CMR
- health subject group (No Intervention): Healthy subjects (30) will be enrolled as controls at baseline.

INTERVENTIONS:
Device: CMR
  Arms: CMR group; Placebo group

SUMMARY:
Magnetic resonance (MR) imaging is a widely used and well-established noninvasive medical diagnostic imaging tool. By using a static and a gradient magnetic field in combination with a radiofrequency field (RF), MR provides excellent contrast among different tissues of the body. Although long-term effects on human health from exposure to strong static magnetic fields seem unlikely, acute effects such as vertigo, nausea, change in blood pressure, reversible arrhythmia, and neurobehavioural effects have been documented from occupational exposition to 1.5 T. Cardiac MR (CMR) imaging requires some of the strongest and fastest switching electromagnetic gradients available in MR exposing the patients to the highest administered energy levels accepted by the controlling authorities. Studies focusing on experimental teratogenic or carcinogenic effects of MR revealed conflicting results. Since CMR is emerging as one of the fastest growing new fields of broad MR application, it is of particular concern that a recent in vitro study with CMR sequences has reported on CMR-induced DNA damages in white blood cells up to 24 h after exposure to 1.5 T CMR. Therefore, we hypothesized that CMR can induce the damage of endothelium and endothelial progenitor cells in type 2 diabetes

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age 30 to 65 years old
* Type 2 diabetes

Exclusion Criteria:

* Renal and liver function dysfunction
* Heart failure
* Malignancy
* Patients with contraindications to cardiac magnetic resonance (CMR)
* Patients with clinical detectable angiopathy

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2013-12; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Changes of endothelium-dependent arterial dilation before and after CMR in type 2 diabetes | 3 days
  The endothelium-dependent arterial dilation was measured at baseline, 1day, 2 day, 3 day after CMR.

SECONDARY OUTCOMES:
Changes of endothelial progenitor cells before and after CMR in peripheral blood | 3 days
  The numbers of endothelial progenitor cells was determined at baseline, 1 day, 2 day, 3 day after CMR.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangda Xiang, Wuhan, Hubei, China

REFERENCES:
- [Derived] Xiang G, Xiang L, He H, Zhang J, Dong J. Impact of cardiac magnetic resonance on endothelial function in type 2 diabetic patients. Atherosclerosis. 2015 Mar;239(1):131-6. doi: 10.1016/j.atherosclerosis.2014.12.028. Epub 2015 Jan 13. PMID 25602854